CLINICAL TRIAL: NCT05221996
Title: Minimal-Dose Resistance Training for Improving sIgA and Cortisol Among Young, Health and Sedentary People
Brief Title: Minimal-Dose Resistance Training for Improving sIgA and Cortisol
Acronym: sIgA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, Luis Berlanga, Principal Investigator, Universidad Francisco de Vitoria
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: UFV2022
Record Dates: First submitted 2022-02-02; First posted 2022-02-03 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Resistance Training; Immune System
Keywords: resistance training; immune system; cortisol
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance exercise for 10 min (Experimental): Resistance circuit training of 10 min
  Interventions: Behavioral: Resistance training
- Resistance exercise for 20 min (Experimental): Resistance circuit training of 20 min
  Interventions: Behavioral: Resistance training
- Resistance exercise for 30 min (Experimental): Resistance circuit training of 30 min
  Interventions: Behavioral: Resistance training

INTERVENTIONS:
Behavioral: Resistance training — Resistance circuit training

SUMMARY:
Whereas the role of endurance training on immune function has been widely studied, little is known about the role of resistance training (RT). In this cross-over randomized controlled study, it will be analysed the effects of three RT protocols which only differs in volume in improving secretory immunoglobulin A (sIgA) and cortisol in saliva among young, health and sedentary people

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years
* Sedentary

Exclusion Criteria:

* to have had COVID-19 during the last 3 months
* to have been vaccinated against COVID-19 during the last 3 months
* physical limitations or health problems

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Concentration of secretory immunoglobulin A (sIgA) | 2 weeks
  Secretory Immunoglobulin A in saliva

SECONDARY OUTCOMES:
Concentration of salivary cortisol (Scortisol) | 2 weeks
  Cortisol in saliva

CONTACTS AND LOCATIONS:
Overall Officials: Luis Berlanga, Principal Investigator — Universidad Francisco de Vitoria
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No